CLINICAL TRIAL: NCT06215924
Title: Investigation of the Effects of Postisometric Relaxation Technique Applied to Pelvic Floor Muscles on Constipation Severity, Quality of Life, Anal Pain, Muscle Function and Sexual Function in Female Patients With Dyssynergic Defecation
Brief Title: The Effects of Postisometric Relaxation Technique in Female Patients With Dyssynergic Defecation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Nuriye BUYUKTAS, Principal Investigator, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nuriye Büyüktaş
Record Dates: First submitted 2023-12-22; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Constipation - Functional; Pelvic Floor Disorders; Pelvic Floor Dyssynergia
Keywords: dyssynergic defecation; functional constipation; pelvic floor physiotherapy; pelvic health; postisometric relaxation technique
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Reverse Kegel' exercise group (Active Comparator): In addition to the training given by the physician, patients will be taught the 'Reverse Kegel' exercise. The 'Reverse Kegel' exercise is an exercise that is used to relax the pelvic floor muscles. To practice the exercise, patients will be asked to lie in a supine position with a support under the knees. In this position, patients will be asked to relax the pelvic floor muscles while breathing through their nose, maintain this movement for 5 seconds, and tighten the pelvic floor muscles while exhaling. Patients will be advised to do this exercise for 5 sets, 10 repetitions during the day. On the day of the training, initial evaluations will be made to the patients before the exercise training is given. Evaluations will be repeated at the end of the second and fourth week.
  Interventions: Other: Reverse Kegel exercise
- 'Postisometric Relaxation Technique' group (Experimental): In addition to training given by the physican, internal digital Postisometric Relaxation method will be applied to the patients in this group from the anal region. Application will be made to the muscles where muscle spasm, movement restriction and pain are detected. The patient will be asked to perform a contraction against the digital resistance with maximum force and maintain this contraction for 5 seconds, actively relax after 5 seconds. During relaxation, stretching will be applied for 30 seconds by digitally supporting the movement of the pelvic floor muscles. The process will be performed with 5 repetitions. The application will be made 2 days a week for 4 weeks. On the day of the training, initial evaluations will be made to the patients before the exercise training is given.Evaluations will be repeated at the end of the second and fourth week.
  Interventions: Other: Postisometric Relaxation Technique

INTERVENTIONS:
Other: Reverse Kegel exercise — In addition to the training given by the physician, patients will be taught the 'Reverse Kegel' exercise. The 'Reverse Kegel' exercise is an exercise that is used to relax the pelvic floor muscles. To practice the exercise, patients will be asked to lie in a supine position with a support under the knees. In this position, patients will be asked to relax the pelvic floor muscles while breathing through their nose, maintain this movement for 5 seconds, and tighten the pelvic floor muscles while exhaling. Patients will be advised to do this exercise for 5 sets, 10 repetitions during the day. On the day of the training, initial evaluations will be made to the patients before the exercise training is given. Evaluations will be repeated at the end of the second and fourth week.
  Arms: 'Reverse Kegel' exercise group
Other: Postisometric Relaxation Technique — In addition to training given by the physican, internal digital Postisometric Relaxation method will be applied to the patients in this group from the anal region. Application will be made to the muscles where muscle spasm, movement restriction and pain are detected. The patient will be asked to perform a contraction against the digital resistance with maximum force and maintain this contraction for 5 seconds, actively relax after 5 seconds. During relaxation, stretching will be applied for 30 seconds by digitally supporting the movement of the pelvic floor muscles. The process will be performed with 5 repetitions. The application will be made 2 days a week for 4 weeks. On the day of the training, initial evaluations will be made to the patients before the exercise training is given.Evaluations will be repeated at the end of the second and fourth week.
  Arms: 'Postisometric Relaxation Technique' group

SUMMARY:
Functional bowel diseases are defined as chronic disorders of the gastrointestinal tract characterized by abdominal pain, bloating, tension and/or defecation abnormalities. Functional bowel diseases are studied under five headings: functional constipation, functional diarrhea, functional abdominal bloating / tightness and unclassifiable functional bowel disorders. Functional constipation is divided into three categories as normal transition-time constipation, slow transition-time constipation and defecation disorders. Defecation disorders occur due to improper use of pelvic floor muscles and anorectal muscles or anatomical abnormalities and account for 1/3 of all constipation. Defecation disorders characterized by excessive straining, incomplete defecation sensation, difficult and painful defecation are defined as narrowing of the fecal exit path due to involuntary pelvic floor contractions or posterior compartment pelvic organ prolapse. Non-pharmacological treatment in the treatment of functional constipation is considered as the first-line treatment and includes information about the nutrition, fiber-liquid consumption, physical activity and toilet training of patients. Biofeedback therapy is often recommended in patients with defecation disorders in the literature, and there are studies showing that it is superior to laxative use and placebo applications in the studies conducted. However, the fact that it is difficult and costly to achieve Biofeedback treatment, the method used allows movement at a certain angle and does not include the stretching method seems to be a disadvantage. Postisometric Relaxation technique is used in cases of pain, muscle spasm and movement limitations. People with defecation disorders experience spasms, pain and movement limitations in the pelvic floor muscles. For this reason, the investigators think that the Postisometric Relaxation technique may be effective in patients with defecation disorders, and it will also provide advantages due to the fact that the method is easily accessible, does not require extra materials and devices, and has a stretching effect. The aim of this study is to investigate the effect of Postisometric Relaxation technique on constipation severity, quality of life, anal pain, muscle function and sexual function in patients with defecation disorder.

ELIGIBILITY:
Inclusion Criteria:

* Being the ages between 18-55
* Being a women
* Having been diagnosed with dyssynergic defecation by a physician
* Not using Laxatives

Exclusion Criteria:

* Having undergone anal region surgery in the last 6 months
* Having had Botox in the last 6 months
* Being in the menopause period
* Having been diagnosed with cancer
* Having a mental problem • Having previously received pelvic floor physiotherapy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female aged between 18-55, female with dyssynergic defecation
Enrollment: 42 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Constipation Severity | Before treatment, end of the second week, end of the fourth week
  The Constipation Severity Scale will be used. It contains a total of 16 questions and is scored between 0-73. High scores indicate that the severity of constipation is excessive.

SECONDARY OUTCOMES:
Quality of Life due to Constipation | Before treatment, end of the second week, end of the fourth week
  The Constipation Quality of life Scale will be used. It contains a total of 28 questions and is scored between 28-140. The high scores obtained from the scale indicate that the quality of life is poor.
Anal Pain | Before treatment, end of the second week, end of the fourth week
  The Visual Analog Scale will be used. In this scale, numbered from 0 to 10, 0 refers to the absence of any pain; 10 refers to the most severe pain.
Sexual Function | Before treatment and end of the fourth week
  The Female Sexual Function Index will be used. The scale contains a total of 19 questions to evaluate sexual functions in the last 4 weeks and is scored between 0-95. High scores obtained from the scale indicate that sexual function is negatively affected.
Function of the pelvic floor muscles | Before treatment, end of the second week, end of the fourth week
  Measurement will be made with a electromyography device (NeuroTrac® MyoPlus Pro). Superficial anal prob will be used. The prob will be inserted rectally to measure the activity of the pelvic floor muscles during contraction and resting. Participants will be asked to contract and relax the pelvic floor muscles for 5 repetitions. The average amount of 5 contraction and relaxation of the measurement will be recorded in micro volts. High resting scores indicate that the pelvic floor muscle can not adequatly relax.

OTHER OUTCOMES:
The impact of Dyssynergic Defecation on other pelvic floor disorders | Before treatment, end of the second week, end of the fourth week
  The Pelvic Floor Impact Questionnaire will be used. It consists of 21 questions and is scored between 0-300. A high score indicates that the degree of complaint of pelvic floor dysfunction is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuriye Büyüktaş, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided